CLINICAL TRIAL: NCT01857869
Title: Efficacy, Safety and Immunogenicity Study of GSK Biologicals' Candidate Malaria Vaccine 257049 in the Sporozoite Challenge Model in Healthy Malaria-naïve Adults
Brief Title: Efficacy, Safety and Immunogenicity Study of GlaxoSmithKline(GSK) Biologicals' Candidate Malaria Vaccine 257049 in the Sporozoite Challenge Model in Healthy Malaria-naïve Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 117014
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Malaria
Keywords: Efficacy; Sporozoite challenge model; Malaria; Immunogenicity; Malaria- naïve adults; Safety
MeSH Terms: conditions — Malaria | interventions — RTS,S-AS01B vaccine

ARMS (3):
- GSK257049-0,1,7M Group (Experimental): Subjects receiving 2 doses of GSK257049 vaccine given at 0 and 1 months and followed 6 months later (At Month 7) by another dose of GSK257049 vaccine.
  Interventions: Biological: GSK257049 Dosage 1
- GSK257049-0,1,2M Group (Experimental): Subjects receiving 3 doses of GSK257049 vaccine given one month apart (0,1 and 2 months).
  Interventions: Biological: GSK257049 Dosage 2
- Infectivity Control Group (Experimental): Volunteers who did not receive any immunization but underwent sporozoite challenge
  Interventions: Procedure: Sporozoite-infected mosquitoes challenge

INTERVENTIONS:
Biological: GSK257049 Dosage 1 — RTS,S/AS01B administered as 0.5 mL dose at 0 and 1 months and 0.1 mL dose at 7 months for 0,1,7 M Group (delayed fractional dose group). In subjects unprotected in the first challenge, to receive a booster with a fractional dose of RTS,S/AS01B followed by rechallenge. In subjects protected in the first challenge, randomization to receive or not receive a booster with a fractional dose of RTS,S/AS01B followed by rechallenge.
  Other Names: S/AS01B; RTS
  Arms: GSK257049-0,1,7M Group
Biological: GSK257049 Dosage 2 — RTS,S/AS01B administered as three doses of 0.5mL given one month apart (0, 1, 2 M group) in the challenge model. In subjects unprotected in the first challenge, to receive a booster with a fractional dose of RTS,S/AS01B followed by rechallenge. In subjects protected in the first challenge, randomization to receive or not receive a booster with a fractional dose of RTS,S/AS01B followed by rechallenge.
  Other Names: RTS; S/AS01B
  Arms: GSK257049-0,1,2M Group
Procedure: Sporozoite-infected mosquitoes challenge — Mosquitoes infected approximately 2-3 weeks earlier that are likely to contain sporozoites in their salivary glands will be allowed to feed on the volunteers. For each volunteer, five mosquitoes will be allowed to feed over five minutes, after which they will be dissected to confirm how many were infected, and the salivary glands scored.
  The challenge is scheduled to occur approximately 21 days (3 weeks) after the last vaccination visit (Study Day 196). Volunteers who reconsent for the boost/rechallenge phase will be rechallenged with sporozoite-infected mosquitoes, scheduled to occur approximately 21 days (3 weeks) after the booster dose (Booster Phase Study Day 21).
  Arms: Infectivity Control Group

SUMMARY:
This study is designed to evaluate safety, reactogenicity, immunogenicity, and efficacy of GSK Biological's malaria candidate vaccine 257049 administered as standard doses at 0 and 1 months and 1/5th standard dose at 7 months (delayed fractional dose group) and 257049 administered as three standard doses one month apart (0, 1, 2-month group) in healthy malaria-naïve volunteers aged 18-50 years in the sporozoite challenge model.

An additional, delayed sporozoite challenge will assess persistence of protection induced by the primary immune schedule and if an additional dose can provide protection in those unprotected by the initial vaccination series.

DETAILED DESCRIPTION:
This protocol posting has been amended to reflect changes in Amendment 1 of the Protocol (20 April 2014).

Rationale for Protocol Amendment 1:

• In order to assess whether protection is maintained over time, and assess boostability, the protocol has been amended to incorporate another sporozoite challenge, after a single boost of 1/5th standard dose of RTS,S/AS01B, or no boost.

Study design:

* Dependent upon enrolment date during the screening period, the study duration will be approximately 19 months for each vaccinated subject in the delayed fractional dose group, 14 months for each vaccinated subject in the 0, 1, 2-month group, 7 months for each infectivity control subject in the challenge phase and 6 months for each infectivity control subject in the rechallenge phase.
* Vaccination schedules:

  * 0, 1, 7-month followed by sporozoite challenge 21 days (3 weeks) after the third vaccination, with subsequent boosting/no boosting at Booster Phase Study Day 0 followed by sporozoite rechallenge 3 weeks post boost/no boost.
  * 0, 1, 2-month followed by sporozoite challenge 21 days (3 weeks) after the third vaccination, with subsequent boosting/no boosting at Booster Phase Study Day 0 followed by sporozoite rechallenge 3 weeks post boost/no boost.
* Safety and immunogenicity will be evaluated during the study up to 3 months after rechallenge (Booster Phase Study Day 105).
* Treatment allocation:

  * Non-randomized for primary phase; subjects will be enrolled to different study groups in a consecutive manner, to ensure the day of sporozoite challenge (conducted over two days) is the same for all.
  * For the booster and rechallenge phase, subjects unprotected during the first challenge will receive a 1/5th RTS,S/AS01B booster dose while subjects from each group who were protected in the first challenge will be randomized to receive a 1/5th RTS,S/AS01B booster dose or no booster dose.

This protocol posting has been amended to reflect changes in Amendment 2 of the Protocol (08 January 2015) Rationale for Protocol Amendment 2: In order to have sufficient blood samples for future assay development or testing, evaluation of Hepatitis B (HBs) cellular-mediated immunogenicity (CMI) was de-prioritised from a secondary outcome measure to a tertiary secondary outcome measure and will only be conducted if sufficient cells are available from the thawn cryotube(s) that will be used for circumsporozoite protein (CS) testing.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for enrolment to the primary phase:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or non-pregnant female 18 to 50 years of age at the time of first vaccination.
* Written informed consent obtained from the subject before screening procedures.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Available to participate for the duration of the study (approximately 15 months per vaccinated subject in the delayed fractional dose group, approximately 10 months per vaccinated subject in the 0, 1, 2-month schedule and approximately 7 months per subject in the infectivity control group).
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate FDA-approved contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate FDA-approved contraception during the entire treatment period and for 2 months after completion of the vaccination series and/or malaria challenge.

Inclusion criteria for enrolment to the booster phase:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject before screening procedures.
* Subjects vaccinated in the primary phase of the study (not applicable to new infectivity controls), having undergone sporozoite challenge during the primary phase of the study.
* Available to participate for the duration of the booster phase of the study (approximately 3 months).
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the booster phase of the study, if the subject:

  * has practiced adequate FDA-approved contraception for 30 days prior to day of booster vaccination, and
  * has a negative pregnancy test on the day of booster vaccination, and
  * has agreed to continue adequate FDA-approved contraception during the entire treatment period and for 2 months after completion of the booster vaccination and/or malaria rechallenge.

Exclusion Criteria:

For enrolment to the primary & booster phase:

* Any confirmed or suspected immunosuppressive or immunodeficient condition, including immunodeficiency virus (HIV) infection.
* Acute disease and/or fever at the time of enrolment to booster phase.

  * Acute disease is defined as the presence of a moderate or severe illness with or without fever. Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
  * Fever is defined as temperature ≥ 38.0°C (100.4°F) on oral, axillary or tympanic setting. The preferred route for recording temperature in this study will be oral.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Evidence of increased cardiovascular disease risk, "moderate" or "high", according to the National health and nutrition examination survey I (NHANES I) criteria.

Note: NHANES I criteria will be applied for all subjects including subjects aged 18-35 years old.

* An abnormal baseline screening electrocardiogram (EKG), defined as one showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm excluding isolated premature atrial contractions; right or left bundle branch block; or advanced A-V heart block.
* Female who intends to become pregnant during the study or planning to discontinue contraceptive measures.

For enrolment to the primary phase:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 7 days of the first dose of vaccines.
* Prior receipt of an investigational malaria vaccine.
* Chronic use of antibiotics with antimalarial effects.
* History of malaria chemoprophylaxis within 60 days prior to vaccination.
* Any history of malaria.
* Planned travel to malaria endemic areas during the study period.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s) including latex.
* History of allergic disease or reactions likely to be exacerbated by chloroquine.
* History of psoriasis and porphyria, which may be exacerbated after chloroquine treatment.
* Current use of medications known to cause drug reactions to chloroquine.
* Any history of anaphylaxis in reaction to any previous vaccination.
* History of severe reactions to mosquito bites.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune modifying drugs within six months prior to first vaccine dose. For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 20 mg/day. Inhaled and topical steroids are allowed.
* Family history of congenital or hereditary immunodeficiency.
* History of splenectomy.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures, except for a single episode of simple febrile seizure in childhood.
* Any abnormal baseline laboratory screening tests: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), creatinine, hemoglobin, platelet count, total white blood cell count, out of normal range as defined in the protocol.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Personal history of autoimmune disease.
* Seropositive for hepatitis B surface antigen or Hepatitis C virus.
* Pregnant or lactating female.
* Suspected or known current alcohol abuse.
* Chronic or active intravenous drug use.
* History of blood donation within 56 days preceding enrolment.
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study.

For enrolment to the booster phase:

* Planned use of any investigational or non-registered product other than the study vaccine during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 7 days of booster dose of study vaccine.
* Planned administration of immunoglobulins and/or any blood products during the study period.
* An abnormal baseline laboratory screening test, graded 2 or more as defined in the protocol.
* Any abnormal baseline laboratory screening tests out of normal range as defined in the protocol and of clinical concern according to the Principal Investigator.
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in the booster phase of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-05-20 (Actual); Primary Completion 2014-03-24 (Actual); Study Completion 2014-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Regules JA, Cicatelli SB, Bennett JW, Paolino KM, Twomey PS, Moon JE, Kathcart AK, Hauns KD, Komisar JL, Qabar AN, Davidson SA, Dutta S, Griffith ME, Magee CD, Wojnarski M, Livezey JR, Kress AT, Waterman PE, Jongert E, Wille-Reece U, Volkmuth W, Emerling D, Robinson WH, Lievens M, Morelle D, Lee CK, Yassin-Rajkumar B, Weltzin R, Cohen J, Paris RM, Waters NC, Birkett AJ, Kaslow DC, Ballou WR, Ockenhouse CF, Vekemans J. Fractional Third and Fourth Dose of RTS,S/AS01 Malaria Candidate Vaccine: A Phase 2a Controlled Human Malaria Parasite Infection and Immunogenicity Study. J Infect Dis. 2016 Sep 1;214(5):762-71. doi: 10.1093/infdis/jiw237. Epub 2016 Jun 13. PMID 27296848
- [Derived] Spreng RL, Seaton KE, Lin L, Hilliard S, Horn GQ, Abraha M, Deal AW, Li K, Carnacchi AJ, Feeney E, Shabbir S, Zhang L, Bekker V, Mudrak SV, Dutta S, Mercer LD, Gregory S, King CR, Wille-Reece U, Jongert E, Kisalu NK, Tomaras GD, Dennison SM. Identification of RTS,S/AS01 vaccine-induced humoral biomarkers predictive of protection against controlled human malaria infection. JCI Insight. 2024 Oct 8;9(19):e178801. doi: 10.1172/jci.insight.178801. PMID 39377226
- [Derived] Oyen D, Torres JL, Wille-Reece U, Ockenhouse CF, Emerling D, Glanville J, Volkmuth W, Flores-Garcia Y, Zavala F, Ward AB, King CR, Wilson IA. Structural basis for antibody recognition of the NANP repeats in Plasmodium falciparum circumsporozoite protein. Proc Natl Acad Sci U S A. 2017 Nov 28;114(48):E10438-E10445. doi: 10.1073/pnas.1715812114. Epub 2017 Nov 14. PMID 29138320
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 117014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 64 subjects originally enrolled in the study, 1 subject was not included in the Intention-to-Treat Cohort. The design of the study included 4 epochs (see pre-assignment details).
Pre-assignment Details: Primary Phase (screening, vaccination [delayed fractional dose group and 0, 1, 2-month group] & challenge): Study Day (D) 217 to D245 - Follow-up: D259 to D376 - Booster (Bst) Phase (re-screening [delayed fractional dose group and 0, 1, 2-month group], vaccination & re-challange): Bst Phase Study D20 to D49 - Follow-up: Bst Phase Study D77 to D105.
Groups:
- GSK257049-0,1,7M Group: Subjects receiving 2 doses of GSK257049 vaccine given at 0 and 1 months and followed 6 months later (At Month 7) by a fractional dose of GSK257049 vaccine and underwent sporozoite challenge (controlled human malaria infection [CHMI]).
- GSK257049-0,1,2M Group: Subjects receiving 3 doses of GSK257049 vaccine given one month apart (0,1 and 2 months) and underwent sporozoite challenge (CHMI).
- Infectivity Control Group: Volunteers who did not receive any immunization but underwent sporozoite challenge (CHMI).
- GSK257049-0,1,7M P-NoBo Group: Subjects from GSK257049-0,1,7M Group who were protected (P) during first CHMI and who received no booster dose (NoBo) of GSK257049 vaccine and underwent sporozoite rechallenge.
- GSK257049-0,1,7M P-Bo Group: Subjects from GSK257049-0,1,7M Group who were protected (P) during first CHMI and who received a booster fractional low-formulated (Bo) of GSK257049 vaccine and underwent sporozoite rechallange.
- GSK257049-0,1,7M NP-Bo Group: Subjects from GSK257049-0,1,7M Group who were not protected (NP) during first CHMI and who received a booster fractional low-formulated (Bo) of GSK257049 vaccine and underwent sporozoite rechallange.
- GSK257049-0,1,2M P-NoBo Group: Subjects from GSK257049-0,1,2M Group who were protected (P) during first CHMI and who received no booster dose (NoBo) of GSK257049 vaccine and underwent sporozoite rechallange.
- GSK257049-0,1,2M P-Bo Group: Subjects from GSK257049-0,1,2M Group who were protected (P) during first CHMI and who received a booster fractional (Bo) of GSK257049 vaccine and underwent sporozoite rechallange.
- GSK257049-0,1,2M NP-Bo Group: Subjects from GSK257049-0,1,2M Group who were not protected (NP) during first CHMI and who received a booster fractional (Bo) of GSK257049 vaccine and underwent sporozoite rechallange.
- Control Group Follow-up: Subjects from Control Group in Primary Phase who remained uninfected with P. falciparum malaria and enrolled as infectivity controls for Follow-up Phase to undergo sporozoite rechallange.
Period: Primary/Challenge Phase
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group | GSK257049-0,1,7M P-NoBo Group | GSK257049-0,1,7M P-Bo Group | GSK257049-0,1,7M NP-Bo Group | GSK257049-0,1,2M P-NoBo Group | GSK257049-0,1,2M P-Bo Group | GSK257049-0,1,2M NP-Bo Group | Control Group Follow-up
Started | 34 | 17 | 12 | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase)
Completed | 29 | 16 | 12 | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase) | 0 (Only GSK257049-0,1,7M,GSK257049-0,1,2M and Infectivity Control Groups were included in Primary phase)
Not Completed | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Booster/Rechallenge Phase
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group | GSK257049-0,1,7M P-NoBo Group | GSK257049-0,1,7M P-Bo Group | GSK257049-0,1,7M NP-Bo Group | GSK257049-0,1,2M P-NoBo Group | GSK257049-0,1,2M P-Bo Group | GSK257049-0,1,2M NP-Bo Group | Control Group Follow-up
Started | 0 (GSK257049-0,1,7M, GSK257049-0,1,2M and Infectivity Control Groups were not included in Booster phase) | 0 (GSK257049-0,1,7M, GSK257049-0,1,2M and Infectivity Control Groups were not included in Booster phase) | 0 (GSK257049-0,1,7M, GSK257049-0,1,2M and Infectivity Control Groups were not included in Booster phase) | 9 | 10 | 2 | 5 | 4 | 3 | 6
Completed | 0 (GSK257049-0,1,7M, GSK257049-0,1,2M and Infectivity Control Groups were not included in Booster phase) | 0 (GSK257049-0,1,7M, GSK257049-0,1,2M and Infectivity Control Groups were not included in Booster phase) | 0 (GSK257049-0,1,7M, GSK257049-0,1,2M and Infectivity Control Groups were not included in Booster phase) | 7 | 10 | 2 | 5 | 4 | 3 | 6
Not Completed | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Volunteer took antibiotic pre-challenge | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants included in the Booster/Rechallenge Phase (0,1,7 M P-NoBo Group; 0,1,7 M P-Bo Group; 0,1,7 NP-Bo Group; 0,1,2 M P-NoBo Group; 0,1,2 M P-Bo Group; 0,1,2 M NP-Bo Group; and Control Group Follow-up) were also in Primary/Challenge Phase (GSK257049-0,1,7M Group; GSK257049-0,1,2M Group; and Infectivity Control Group).
Groups:
- GSK257049-0,1,7M Group: Subjects receiving 2 doses of GSK257049 vaccine given at 0 and 1 months and followed 6 months later (At Month 7) by a fractional dose of GSK257049 vaccine and underwent sporozoite challenge (CHMI).
- GSK257049-0,1,2M P-Bo Group: Subjects from GSK257049-0,1,2M Group who were protected (P) during first CHMI and who received a booster fractional low-formulated (Bo) of GSK257049 vaccine and underwent sporozoite rechallange.
- GSK257049-0,1,2M NP-Bo Group: Subjects from GSK257049-0,1,2M Group who were not protected (NP) during first CHMI and who received a booster fractional low-formulated (Bo) of GSK257049 vaccine and underwent sporozoite rechallange.
- Total: Total of all reporting groups
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group | GSK257049-0,1,7M P-NoBo Group | GSK257049-0,1,7M P-Bo Group | GSK257049-0,1,7M NP-Bo Group | GSK257049-0,1,2M P-NoBo Group | GSK257049-0,1,2M P-Bo Group | GSK257049-0,1,2M NP-Bo Group | Control Group Follow-up | Total
Number analyzed (Participants) | 34 | 17 | 12 | 7 | 10 | 2 | 5 | 4 | 3 | 6 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: This baseline measure refers to the Primary/challenge phase population.
  Years
    number analyzed (Participants) | 34 | 17 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63
    (all) | 34.4 (8.6) | 30.1 (7.9) | 36.4 (8.7) |  |  |  |  |  |  |  | 33.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This baseline measure refers to the Primary/challenge phase population.
  Participants
    number analyzed (Participants) | 34 | 17 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63
    Female | 15 | 6 | 7 |  |  |  |  |  |  |  | 28
    Male | 19 | 11 | 5 |  |  |  |  |  |  |  | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: This baseline measure refers to the Primary/challenge phase population.
  Participants
    Geographic ancestry: number analyzed (Participants) | 34 | 17 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63
    Geographic ancestry: African Heritage/African American | 15 | 5 | 5 |  |  |  |  |  |  |  | 25
    Geographic ancestry: Asian - Central/South Asian Heritage | 1 | 0 | 0 |  |  |  |  |  |  |  | 1
    Geographic ancestry: Asian - South East Asian Heritage | 2 | 0 | 0 |  |  |  |  |  |  |  | 2
    Geographic ancestry: White - Caucasian/European Heritage | 13 | 10 | 5 |  |  |  |  |  |  |  | 28
    Geographic ancestry: Unspecified | 3 | 2 | 2 |  |  |  |  |  |  |  | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Plasmodium Falciparum Parasitemia Defined by a Positive Blood Slide, Following Sporozoite Challenge
Description: The definition of malaria for primary and secondary efficacy outcomes is the appearance of asexual blood stage P. falciparum parasites detected by blood slide at any time post challenge/rechallenge up to 28 days.
Time Frame: 28 days post-challenge (Study Day 245)
Population: The analysis was based on the According-to-Protocol (ATP) population for immunogenicity and efficacy, which included all subjects who complied with the protocol requirements and underwent P. falciparum CHMI.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 30 | 16 | 12
Participants | 4 | 6 | 12
Statistical Analysis 1: Comparison: GSK257049-0,1,7M Group vs Infectivity Control Group; Vaccine efficacy (VE) was defined as 100*(1-Relative Risk [RR]); Test type: Other; p < 0.0001, Mantel Haenszel — Two-sided Fisher Exact test was used for the comparison of malaria incidence after first/second CHMI between the compared groups; 1-Relative Risk = 86.7, 95% CI 2-sided [66.8 to 94.6]
Statistical Analysis 2: Comparison: GSK257049-0,1,2M Group vs Infectivity Control Group; Vaccine efficacy (VE) was defined as 100*(1-Relative Risk [RR]); Test type: Other; p = 0.0009, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; 1-Relative Risk = 62.5, 95% CI 2-sided [29.4 to 80.1]

2. Secondary Outcome: Time to Onset of P. Falciparum Parasitemia Infection Defined by a Positive Blood Slide, Following Sporozoite Challenge
Description: The time to onset was expressed in days. The definition of malaria infection for primary and secondary efficacy outcomes is the appearance of asexual blood stage P. falciparum parasites detected by blood slide at any time post challenge/rechallenge up to 28 days.
Time Frame: Up to 28 days post-challenge (Study Day 245)
Population: The analysis was based on the ATP population for immunogenicity and efficacy, which included all subjects who complied with the protocol requirements and underwent P. falciparum CHMI. This analysis included those subjects with a positive blood slide.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 4 | 6 | 12
Days | 17 (6) | 15 (5) | 13 (1)

3. Secondary Outcome: Number of Subjects With Plasmodium Falciparum Parasitemia Defined by a Positive Blood Slide, Following Sporozoite Rechallenge
Description: The definition of malaria infection for primary and secondary efficacy outcomes is the appearance of asexual blood stage P. falciparum parasites detected by blood slide at any time post challenge/rechallenge up to 28 days.
Time Frame: Up to 28 days post rechallenge (Booster Phase Day 49)
Population: The analysis was based on the ATP population for immunogenicity and efficacy for the rechallenge Phase, which included all subjects from the ATP population for immunogenicity and efficacy who consented to the rechallenge.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049-0,1,7M P-NoBo Group | GSK257049-0,1,7M P-Bo Group | GSK257049-0,1,7M NP-Bo Group | GSK257049-0,1,2M P-NoBo Group | GSK257049-0,1,2M P-Bo Group | GSK257049-0,1,2M NP-Bo Group | Control Group Follow-up
Number analyzed (Participants) | 7 | 10 | 2 | 5 | 4 | 3 | 6
Participants | 4 | 1 | 0 | 4 | 3 | 1 | 6

4. Secondary Outcome: Time to Onset of P. Falciparum Parasitemia Infection Defined by a Positive Blood Slide, Following Sporozoite Rechallenge
Description: as for outcome 2
Time Frame: Up to 28 days post rechallenge (Booster Phase Day 49)
Population: The analysis was based on the ATP population for immunogenicity and efficacy for the rechallenge Phase, which included all subjects from the ATP population for immunogenicity and efficacy who consented to the rechallenge. This analysis included those subjects with a positive blood slide.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK257049-0,1,7M P-NoBo Group | GSK257049-0,1,7M P-Bo Group | GSK257049-0,1,2M P-NoBo Group | GSK257049-0,1,2M P-Bo Group | GSK257049-0,1,2M NP-Bo Group | Control Group Follow-up
Number analyzed (Participants) | 4 | 1 | 4 | 3 | 1 | 6
Days | 14 (1) | 14 (0) | 15 (1) | 14 (2) | 14 (0) | 12 (1)

5. Secondary Outcome: Anti-circumsporozoite (Anti-CS) Repeat Region Antibody Concentrations
Description: Anti-CS antibody concentrations were determined by Enzyme Linked Immunosorbent Assay (ELISA) and expressed as EU/mL.
Time Frame: 7 days before vaccination (D-7), post-dose 1 at Day 28, post-dose 2 at Days 42, 56, 98, 196, at DoC Primary Phase (PP) (Day of CHMI = Day 217), at DoC PP (Day 217) + 7, 14, 28, 42, 56, 70, 84, 159 days (Days 224, 231, 245, 259, 273, 287, 301, 376).
Population: The analysis was based on the ATP population for immunogenicity and efficacy, which included all subjects who complied with the protocol requirements and underwent P. falciparum CHMI.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 30 | 16 | 12
EU/mL
  7 days before vaccination: number analyzed (Participants) | 30 | 16 | 0
  7 days before vaccination | 0.3 [0.2 to 0.3] | 0.3 [0.3 to 0.3] |
  At Day 28: number analyzed (Participants) | 29 | 16 | 0
  At Day 28 | 13.1 [6.9 to 25.1] | 16.3 [8.0 to 33.2] |
  At Day 42: number analyzed (Participants) | 28 | 16 | 0
  At Day 42 | 104.2 [76.0 to 142.7] | 64.4 [34.1 to 121.8] |
  At Day 56: number analyzed (Participants) | 29 | 16 | 0
  At Day 56 | 83.3 [59.1 to 117.5] | 57.9 [30.7 to 109.4] |
  At Day 98: number analyzed (Participants) | 28 | 0 | 0
  At Day 98 | 46.1 [30.4 to 69.7] |  |
  At Day 196: number analyzed (Participants) | 30 | 0 | 0
  At Day 196 | 18.3 [11.3 to 29.6] |  |
  At DoC PP (Day 217) | 75.2 [57.8 to 97.8] | 100.1 [63.5 to 157.8] | 0.4 [0.2 to 0.8]
  Day 7 after DoC PP (Day 217) | 75.7 [57.3 to 100.0] | 91.7 [57.5 to 146.2] | 0.4 [0.2 to 0.8]
  Day 14 after DoC PP (Day 217) | 68.9 [51.8 to 91.6] | 79.4 [48.5 to 130.0] | 0.4 [0.2 to 0.8]
  Day 28 after DoC PP (Day 217) | 63.8 [46.8 to 87.0] | 75.7 [45.8 to 125.2] | 0.5 [0.3 to 1.0]
  Day 42 after DoC PP (Day 217) | 57.6 [42.3 to 78.5] | 73.6 [45.3 to 119.7] | 0.6 [0.3 to 1.1]
  Day 56 after DoC PP (Day 217): number analyzed (Participants) | 30 | 14 | 12
  Day 56 after DoC PP (Day 217) | 54.0 [38.9 to 75.0] | 63.2 [34.9 to 114.3] | 0.5 [0.3 to 1.0]
  Day 70 after DoC PP (Day 217): number analyzed (Participants) | 29 | 15 | 12
  Day 70 after DoC PP (Day 217) | 46.9 [33.0 to 66.5] | 59.2 [35.1 to 99.8] | 0.5 [0.3 to 1.0]
  Day 84 after DoC PP (Day 217) | 45.6 [32.1 to 64.8] | 55.3 [34.4 to 88.9] | 0.5 [0.3 to 1.0]
  Day 159 after DoC PP (Day 217): number analyzed (Participants) | 29 | 16 | 12
  Day 159 after DoC PP (Day 217) | 32.8 [22.1 to 48.6] | 34.6 [20.9 to 57.0] | 0.5 [0.3 to 1.0]

6. Secondary Outcome: Anti-CS Repeat Region Antibody Concentrations for the Rechallenge Phase
Description: Anti-CS antibody concentrations were determined by Enzyme Linked Immunosorbent Assay (ELISA) and expressed as EU/mL.
Time Frame: At Day 0 of rechallenge (pre-booster dose) and at DoC PP (Day 217 = Day of rechallenge)
Population: The analysis was based on the ATP population for immunogenicity and efficacy for the rechallenge, which included all subjects from the ATP population for immunogenicity and efficacy who consented to the rechallenge.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | GSK257049-0,1,7M P-NoBo Group | GSK257049-0,1,7M P-Bo Group | GSK257049-0,1,7M NP-Bo Group | GSK257049-0,1,2M P-NoBo Group | GSK257049-0,1,2M P-Bo Group | GSK257049-0,1,2M NP-Bo Group | Control Group Follow-up
Number analyzed (Participants) | 7 | 10 | 2 | 5 | 4 | 3 | 6
EU/mL
  At Day 0 of rechallenge: number analyzed (Participants) | 0 | 10 | 2 | 0 | 4 | 3 | 0
  At Day 0 of rechallenge |  | 30.7 [13.0 to 72.1] | 7.2 [0.0 to 44283115] |  | 35.9 [15.8 to 81.7] | 24.5 [1.8 to 334.0] |
  At DoC PP (Day 217) | 25.7 [10.3 to 64.5] | 86.6 [52.0 to 144.1] | 81.2 [0.0 to 660120.7] | 39.2 [17.2 to 89.4] | 61.7 [13.0 to 292.4] | 53.5 [12.3 to 231.6] | 0.3 [0.2 to 0.4]

7. Secondary Outcome: Frequency of CS Repeat and T-cell Epitope (RT)-Specific Cluster of Differentiation 4 (CD4) T-cells
Description: Frequency of Cluster of Differentiation 4 (CD4) polypositives T-cells with at least 2 cytokines/activation markers between CD40-Ligand (CD40-L), interferon gamma (INF-g), interleukin-2 (IL-2) and tumor necrosis factor-alpha (TNF-a) was assessed for peripheral blood mononuclear cells (PBMC) with intracellular cytokine staining (ICS).
Time Frame: 7 days before vaccination (D-7), post-dose 1 at Day 14, post-dose 2 at Day 42, at DoC PP (Day of CHMI = Day 217), at DoC PP (Day 217) + 7, 28, 84, 159 days (Days 224, 245, 301, 376).
Population: The analysis was based on the ATP population for immunogenicity and efficacy, which included all subjects who complied with the protocol requirements and underwent P. falciparum CHMI, with cellular mediated immunity data available.
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/million CD4 T-cells
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 29 | 16 | 12
CD4+ T-cells/million CD4 T-cells
  7 days before vaccination: number analyzed (Participants) | 29 | 16 | 0
  7 days before vaccination | 61.38 (95.16) | 83.31 (79.40) |
  At Day 14: number analyzed (Participants) | 28 | 15 | 0
  At Day 14 | 168.89 (205.87) | 242.53 (262.97) |
  At Day 42: number analyzed (Participants) | 27 | 15 | 0
  At Day 42 | 1306.11 (1962.03) | 866.87 (779.25) |
  At DoC PP (Day 217): number analyzed (Participants) | 27 | 14 | 12
  At DoC PP (Day 217) | 596.15 (636.60) | 555.86 (487.16) | 57.17 (102.19)
  Day 7 after DoC PP (Day 217): number analyzed (Participants) | 28 | 15 | 12
  Day 7 after DoC PP (Day 217) | 661.61 (711.86) | 539.40 (416.68) | 39.25 (42.40)
  Day 28 after DoC PP (Day 217): number analyzed (Participants) | 28 | 16 | 9
  Day 28 after DoC PP (Day 217) | 626.29 (586.16) | 472.63 (287.64) | 162.22 (275.51)
  Day 84 after DoC PP (Day 217): number analyzed (Participants) | 27 | 13 | 12
  Day 84 after DoC PP (Day 217) | 481.44 (392.44) | 472.63 (287.64) | 90.67 (121.47)
  Day 159 after DoC PP (Day 217): number analyzed (Participants) | 27 | 15 | 11
  Day 159 after DoC PP (Day 217) | 490.00 (401.39) | 307.87 (231.91) | 32.55 (51.06)

8. Secondary Outcome: Frequency of CS Repeat and T-cell Epitope (RT)-Specific CD8 T-cells
Description: Frequency of CD8 polypositives T-cells with at least 2 cytokines/activation markers between CD40-L, INF-g, IL-2 and TNF-a was assessed for PBMC with ICS.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: CD8+ T-cells/million CD8 T-cells
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 29 | 16 | 12
CD8+ T-cells/million CD8 T-cells
  7 days before vaccination: number analyzed (Participants) | 29 | 16 | 0
  7 days before vaccination | 14.10 (20.60) | 9.56 (15.31) |
  At Day 14: number analyzed (Participants) | 28 | 15 | 0
  At Day 14 | 24.61 (43.01) | 17.20 (30.03) |
  At Day 42: number analyzed (Participants) | 27 | 15 | 0
  At Day 42 | 18.7 (46.69) | 27.60 (40.40) |
  At DoC PP (Day 217): number analyzed (Participants) | 27 | 14 | 12
  At DoC PP (Day 217) | 32.52 (57.64) | 28.86 (28.73) | 15.33 (29.06)
  Day 7 after DoC PP (Day 217): number analyzed (Participants) | 28 | 15 | 12
  Day 7 after DoC PP (Day 217) | 19.54 (42.55) | 32.07 (56.77) | 32.00 (53.81)
  Day 28 after DoC PP (Day 217): number analyzed (Participants) | 28 | 16 | 9
  Day 28 after DoC PP (Day 217) | 19.96 (27.35) | 34.81 (66.56) | 17.67 (36.31)
  Day 84 after DoC PP (Day 217): number analyzed (Participants) | 27 | 13 | 12
  Day 84 after DoC PP (Day 217) | 19.89 (54.19) | 20.23 (26.25) | 12.17 (22.91)
  Day 159 after DoC PP (Day 217): number analyzed (Participants) | 27 | 15 | 11
  Day 159 after DoC PP (Day 217) | 26.74 (52.22) | 24.40 (44.30) | 22.00 (33.01)

9. Secondary Outcome: Antibody Concentrations Against Hepatitis B Surface Antigen (Anti-HBs)
Description: Anti-HBs antibody concentrations were determined by Chemiluminometric Immunoassay (CLIA) and expressed as miliinternation units per mililier (mIU/mL).
Time Frame: 7 days before vaccination (D-7), post-dose 1 at Day 28, post-dose 2 at Days 42, 56, 98, 196 after first dose, at DoC PP (Day of CHMI = Day 217), at DoC PP (Day 217)+ 7, 14, 28, 42, 56, 70, 84, 159 days (Days 224, 231, 245, 259, 273, 287, 301, 376).
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 30 | 16 | 12
mIU/mL
  7 days before vaccination: number analyzed (Participants) | 30 | 16 | 0
  7 days before vaccination | 27.5 [11.4 to 66.0] | 28.5 [7.1 to 113.9] |
  At Day 28: number analyzed (Participants) | 29 | 16 | 0
  At Day 28 | 7223.0 [1437.5 to 36292.7] | 7318.2 [643.5 to 83221.5] |
  At Day 42: number analyzed (Participants) | 26 | 16 | 0
  At Day 42 | 35016.9 [14549.0 to 84279.4] | 27205.5 [5504.0 to 134473.9] |
  At Day 56: number analyzed (Participants) | 28 | 16 | 0
  At Day 56 | 21013.0 [8181.7 to 53967.5] | 20625.8 [3809.7 to 111668.5] |
  At Day 98: number analyzed (Participants) | 26 | 0 | 0
  At Day 98 | 12367.7 [5159.9 to 29643.9] |  |
  At Day 196: number analyzed (Participants) | 29 | 0 | 0
  At Day 196 | 9917.0 [4447.7 to 22111.9] |  |
  At DoC PP (Day 217) | 33715.4 [20777.5 to 54709.5] | 31798.7 [8809.6 to 114779.3] | 27.9 [6.6 to 118.1]
  Day 7 after DoC PP (Day 217): number analyzed (Participants) | 30 | 15 | 11
  Day 7 after DoC PP (Day 217) | 29902.6 [18090.1 to 49428.5] | 28989.2 [7097.6 to 118403.1] | 32.5 [7.3 to 145.1]
  Day 14 after DoC PP (Day 217): number analyzed (Participants) | 24 | 15 | 12
  Day 14 after DoC PP (Day 217) | 35401.1 [20513.7 to 61092.8] | 24952.2 [6402.7 to 97242.0] | 25.7 [6.4 to 103.0]
  Day 28 after DoC PP (Day 217): number analyzed (Participants) | 27 | 16 | 12
  Day 28 after DoC PP (Day 217) | 25553.8 [14413.9 to 45303.2] | 25944.1 [7496.3 to 89790.9] | 27.5 [6.5 to 116.4]
  Day 42 after DoC PP (Day 217): number analyzed (Participants) | 26 | 14 | 11
  Day 42 after DoC PP (Day 217) | 23757.6 [13130.3 to 42986.3] | 20000.3 [5110.6 to 78271.6] | 32.8 [7.3 to 146.6]
  Day 56 after DoC PP (Day 217): number analyzed (Participants) | 26 | 13 | 11
  Day 56 after DoC PP (Day 217) | 25917.3 [14012.2 to 47937.4] | 23199.5 [5472.8 to 98343.4] | 34.6 [7.7 to 155.2]
  Day 70 after DoC PP (Day 217): number analyzed (Participants) | 23 | 14 | 11
  Day 70 after DoC PP (Day 217) | 23722.4 [12431.5 to 45268.1] | 23313.8 [6098.3 to 89128.6] | 31.9 [7.3 to 139.8]
  Day 84 after DoC PP (Day 217): number analyzed (Participants) | 29 | 16 | 12
  Day 84 after DoC PP (Day 217) | 19155.1 [10713.8 to 34247.0] | 19631.5 [6184.8 to 62313.2] | 26.3 [6.5 to 106.5]
  Day 159 after DoC PP (Day 217): number analyzed (Participants) | 29 | 16 | 12
  Day 159 after DoC PP (Day 217) | 14459.9 [7702.5 to 27145.8] | 13495.2 [3956.7 to 46028.2] | 26.2 [6.5 to 106.0]

10. Secondary Outcome: Anti-HBs Antibody Concentrations for Rechallenge Phase
Description: Anti-HBs antibody concentrations were determined by Chemiluminometric Immunoassay (CLIA).
Time Frame: At Day 0 of rechallenge (pre-booster dose) and at DoC PP (Day 217 = Day of rechallenge)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK257049-0,1,7M P-NoBo Group | GSK257049-0,1,7M P-Bo Group | GSK257049-0,1,7M NP-Bo Group | GSK257049-0,1,2M P-NoBo Group | GSK257049-0,1,2M P-Bo Group | GSK257049-0,1,2M NP-Bo Group | Control Group Follow-up
Number analyzed (Participants) | 7 | 10 | 2 | 5 | 4 | 3 | 6
mIU/mL
  At Day 9 of rechallenge: number analyzed (Participants) | 0 | 10 | 2 | 0 | 4 | 3 | 0
  At Day 9 of rechallenge |  | 9270.9 [3019.1 to 28468.3] | 6928.3 [0.0 to 280600000000000] |  | 23259.5 [5399.6 to 100192.6] | 15620.0 [268.0 to 910369.4] |
  At DoC PP (Day 217): number analyzed (Participants) | 7 | 9 | 2 | 5 | 4 | 3 | 6
  At DoC PP (Day 217) | 19592.4 [5063.3 to 75812.3] | 24261.5 [10414.9 to 56517.5] | 36809.8 [0.0 to 631600000000] | 6051.9 [340.9 to 107425.7] | 38175.5 [12828.4 to 113604.9] | 34470.4 [6909.0 to 171979.3] | 35.7 [3.8 to 335.7]

11. Secondary Outcome: Anti-CS Repeat Region Immunoglobulin G (IgG) Avidity Index for the Challenge Phase
Description: The avidity index percentage was calculated by anti-CS repeat region concentration under chaotropic reagent/anti-CS repeat region concentration without chaotropic reagent. The median and inter-quartile (Q1 and Q3) range was reported at the prespecified time-points.
Time Frame: Post-dose 1 at Day 28, post-dose 2 at Days 56, and 196, DoC PP (DoC = the day of CHMI, Day 217), DoC PP (Day 217) + 84 days (Day 301) and DoC PP (Day 217) +159 days (Day 376)
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Avidity index
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 30 | 16 | 2
Avidity index
  At Day 28: number analyzed (Participants) | 26 | 15 | 0
  At Day 28 | 25.65 [16.30 to 40.50] | 17.90 [8.30 to 27.80] |
  At Day 56: number analyzed (Participants) | 29 | 16 | 0
  At Day 56 | 37.40 [28.50 to 45.10] | 31.10 [19.85 to 33.50] |
  At Day 196: number analyzed (Participants) | 30 | 0 | 0
  At Day 196 | 28.10 [19.40 to 40.10] |  |
  At DoC PP (Day 217): number analyzed (Participants) | 30 | 16 | 0
  At DoC PP (Day 217) | 40.40 [31.80 to 49.60] | 29.00 [22.40 to 34.05] |
  Day 84 after DoC PP (Day 217): number analyzed (Participants) | 30 | 15 | 2
  Day 84 after DoC PP (Day 217) | 37.40 [32.50 to 44.00] | 28.30 [18.70 to 31.50] | 32.10 [20.50 to 43.70]
  Day 159 after DoC PP (Day 217): number analyzed (Participants) | 29 | 15 | 2
  Day 159 after DoC PP (Day 217) | 36.10 [30.60 to 43.80] | 28.90 [19.60 to 32.70] | 32.05 [21.90 to 42.20]

12. Secondary Outcome: Anti-CS Repeat Region IgG Avidity Index for the Rechallenge Phase
Description: The avidity index percentage was calculated by anti-CS repeat region titer under chaotropic reagent/anti-CS repeat region titer without chaotropic reagent. The median and inter-quartile (Q1 and Q3) range was reported at the prespecified time-points.
Time Frame: Pre-booster dose (Booster phase Day 0) and at DoC Booster/rechallenge phase (Day of Controlled Human Malaria Infection - Day 21)
Population: The analysis was based on the ATP population for immunogenicity and efficacy for the rechallenge, which included all subjects from the ATP population for immunogenicity and efficacy who consented to the rechallenge. Results were not reported for the Control Group Follow-up, since subjects from this group did not receive any immunization.
Measure: Median (Inter-Quartile Range); unit: Avidity index
Arm/Group | GSK257049-0,1,7M P-NoBo Group | GSK257049-0,1,7M P-Bo Group | GSK257049-0,1,7M NP-Bo Group | GSK257049-0,1,2M P-NoBo Group | GSK257049-0,1,2M P-Bo Group | GSK257049-0,1,2M NP-Bo Group
Number analyzed (Participants) | 7 | 10 | 2 | 5 | 4 | 3
Avidity index
  Pre-booster dose: number analyzed (Participants) | 0 | 10 | 2 | 0 | 4 | 3
  Pre-booster dose |  | 41.15 [27.10 to 48.40] | 43.30 [38.60 to 48.00] |  | 21.25 [12.95 to 32.05] | 30.40 [15.50 to 34.70]
  DoC Booster/rechallenge phase (Day 21) | 35.00 [30.40 to 44.10] | 46.55 [44.60 to 51.80] | 50.60 [44.70 to 56.50] | 31.30 [22.80 to 38.60] | 36.80 [21.80 to 39.65] | 31.20 [23.20 to 40.90]

13. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = significant pain at rest, that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was based on the Intention-to-Treat (ITT) population, which included all subjects with at least one vaccine administration documented, who had their symptom sheets filled in. Results were not reported for the Infectivity Control Group, since subjects from this group did not receive any immunization.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group
Number analyzed (Participants) | 34 | 17
Participants
  Any Pain, Dose 1 | 30 | 16
  Grade 3 Pain, Dose 1 | 0 | 0
  Any Redness, Dose 1 | 7 | 8
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 8 | 1
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 33 | 16
  Any Pain, Dose 2 | 28 | 13
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 33 | 16
  Grade 3 Pain, Dose 2 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 33 | 16
  Any Redness, Dose 2 | 13 | 6
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 33 | 16
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 33 | 16
  Any Swelling, Dose 2 | 10 | 2
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 33 | 16
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 30 | 16
  Any Pain, Dose 3 | 21 | 12
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 30 | 16
  Grade 3 Pain, Dose 3 | 0 | 0
  Any Redness, Dose 3: number analyzed (Participants) | 30 | 16
  Any Redness, Dose 3 | 23 | 7
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 30 | 16
  Grade 3 Redness, Dose 3 | 0 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 30 | 16
  Any Swelling, Dose 3 | 17 | 3
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 30 | 16
  Grade 3 Swelling, Dose 3 | 0 | 0
  Any Pain, Across doses | 32 | 16
  Grade 3 Pain, Across doses | 0 | 0
  Any Redness, Across doses | 26 | 12
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 21 | 4
  Grade 3 Swelling, Across doses | 0 | 0

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (nausea, vomiting and/or abdominal pain), headache and fever [defined as axillary temperature equal to or above (≥) 38.0 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was based on the ITT population, which included all subjects with at least one vaccine administration documented, who had their symptom sheets filled in. Results were not reported for the Infectivity Control Group, since subjects from this group did not receive any immunization.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group
Number analyzed (Participants) | 34 | 17
Participants
  Any Fatigue, Dose 1 | 10 | 3
  Related Fatigue, Dose 1 | 9 | 3
  Grade 3 Fatigue, Dose 1 | 1 | 0
  Any Gastrointestinal symptoms, Dose 1 | 4 | 2
  Related Gastrointestinal symptoms, Dose 1 | 4 | 2
  Grade 3 Gastrointestinal symptoms, Dose 1 | 0 | 0
  Any Headache, Dose 1 | 9 | 9
  Related Headache, Dose 1 | 8 | 9
  Grade 3 Headache, Dose 1 | 1 | 0
  Any Temperature, Dose 1 | 3 | 3
  Related Temperature, Dose 1 | 3 | 0
  Grade 3 Temperature, Dose 1 | 0 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 33 | 16
  Any Fatigue, Dose 2 | 15 | 5
  Related Fatigue, Dose 2: number analyzed (Participants) | 33 | 16
  Related Fatigue, Dose 2 | 15 | 5
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 33 | 16
  Grade 3 Fatigue, Dose 2 | 1 | 0
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 33 | 16
  Any Gastrointestinal symptoms, Dose 2 | 3 | 5
  Related Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 33 | 16
  Related Gastrointestinal symptoms, Dose 2 | 3 | 5
  Grade 3 Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 33 | 16
  Grade 3 Gastrointestinal symptoms, Dose 2 | 0 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 33 | 16
  Any Headache, Dose 2 | 15 | 9
  Related Headache, Dose 2: number analyzed (Participants) | 33 | 16
  Related Headache, Dose 2 | 15 | 8
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 33 | 16
  Grade 3 Headache, Dose 2 | 0 | 0
  Any Temperature, Dose 2: number analyzed (Participants) | 33 | 16
  Any Temperature, Dose 2 | 6 | 1
  Related Temperature, Dose 2: number analyzed (Participants) | 33 | 16
  Related Temperature, Dose 2 | 6 | 1
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 33 | 16
  Grade 3 Temperature, Dose 2 | 3 | 0
  Any Fatigue, Dose 3: number analyzed (Participants) | 30 | 16
  Any Fatigue, Dose 3 | 8 | 7
  Related Fatigue, Dose 3: number analyzed (Participants) | 30 | 16
  Related Fatigue, Dose 3 | 8 | 6
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 30 | 16
  Grade 3 Fatigue, Dose 3 | 0 | 0
  Any Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 30 | 16
  Any Gastrointestinal symptoms, Dose 3 | 6 | 2
  Related Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 30 | 16
  Related Gastrointestinal symptoms, Dose 3 | 3 | 2
  Grade 3 Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 30 | 16
  Grade 3 Gastrointestinal symptoms, Dose 3 | 0 | 0
  Any Headache, Dose 3: number analyzed (Participants) | 30 | 16
  Any Headache, Dose 3 | 9 | 6
  Related Headache, Dose 3: number analyzed (Participants) | 30 | 16
  Related Headache, Dose 3 | 7 | 6
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 30 | 16
  Grade 3 Headache, Dose 3 | 0 | 0
  Any Temperature, Dose 3: number analyzed (Participants) | 30 | 16
  Any Temperature, Dose 3 | 0 | 0
  Related Temperature, Dose 3: number analyzed (Participants) | 30 | 16
  Related Temperature, Dose 3 | 0 | 0
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 30 | 16
  Grade 3 Temperature, Dose 3 | 0 | 0
  Any Fatigue, Across doses | 18 | 9
  Related Fatigue, Across doses | 18 | 8
  Grade 3 Fatigue, Across doses | 2 | 0
  Any Gastrointestinal symptoms, Across doses | 7 | 5
  Related Gastrointestinal symptoms, Across doses | 7 | 5
  Grade 3 Gastrointestinal symptoms, Across doses | 0 | 0
  Any Headache, Across doses | 18 | 11
  Related Headache, Across doses | 18 | 11
  Grade 3 Headache, Across doses | 1 | 0
  Any Temperature, Across doses | 8 | 4
  Related Temperature, Across doses | 8 | 1
  Grade 3 Temperature, Across doses | 3 | 0

15. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within the 7-day (Days 0-6) post- booster vaccination period
Population: The analysis was based on the ITT population for the rechallenge, which included subjects from the ITT population consenting to the rechallenge. For the purpose of the analysis, subjects who received a low fractional formulation booster dose of GSK257049 vaccine have been pooled into a single group and results were tabulated accordingly.
Measure: Count of Participants; unit: Participants
Groups:
- Boosted Group: Pooled group comprising subjects from the GSK257049-0,1,7M P-Bo Group; GSK257049-0,1,7M NP-Bo Group; GSK257049-0,1,2M P-Bo Group and GSK257049-0,1,2M NP-Bo Group (protected and not protected subjects from the Primary Phase groups, that received a low fractional formulation booster dose of GSK257049 vaccine).
Arm/Group | Boosted Group
Number analyzed (Participants) | 19
Participants
  Any Pain | 11
  Grade 3 Pain | 0
  Any Redness | 8
  Grade 3 Redness | 0
  Any Swelling | 4
  Grade 3 Swelling | 0

16. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache and fever [defined as axillary temperature equal to or above (≥) 38.0 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 7-day (Days 0-6) post- booster vaccination period
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Boosted Group
Number analyzed (Participants) | 19
Participants
  Any Fatigue | 8
  Related Fatigue | 5
  Grade 3 Fatigue | 0
  Any Gastrointestinal symptoms | 4
  Related Gastrointestinal symptoms | 3
  Grade 3 Gastrointestinal symptoms | 0
  Any Headache | 8
  Related Headache | 6
  Grade 3 Headache | 1
  Any Temperature | 0
  Related Temperature | 0
  Grade 3 Temperature | 0

17. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 30-days (Days 0-29) post-primary vaccination
Population: The analysis was based on the ITT population, which included all subjects with at least one vaccine administration documented. Results were not reported for the Infectivity Control Group, since subjects from this group did not receive any immunization.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group
Number analyzed (Participants) | 34 | 17
Participants | 25 | 16

18. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 17
Time Frame: Within 30-days (Days 0-29) post- booster vaccination
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Boosted Group
Number analyzed (Participants) | 19
Participants | 10

19. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 17
Time Frame: Within 30-days (Days 0-29) post-first CHMI
Population: The analysis was based on the ITT population, which included all subjects with at least one vaccine administration documented and who had post-first CHMI available results.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 30 | 16 | 12
Participants | 25 | 13 | 12

20. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: as for outcome 17
Time Frame: Within 30-days (Days 0-29) post- second CHMI
Population: The analysis was based on the ITT population for the rechallenge, which included subjects from the ITT population consenting to the rechallenge.
Measure: Count of Participants; unit: Participants
Groups:
- Non Boosted Group: Pooled group comprising subjects from the GSK257049-0,1,7M P-NoBo and GSK257049-0,1,2M P-NoBo Group (protected subjects from the Primary Phase groups, that did not receive a booster dose of GSK257049 vaccine.
- Control Group Follow-up: Subjects from Control Group in Primary Phase who remained uninfected with P. falciparum malaria and enrolled as infectivity controls for Follow-up Phase.
Arm/Group | Non Boosted Group | Boosted Group | Control Group Follow-up
Number analyzed (Participants) | 12 | 19 | 6
Participants | 11 | 15 | 6

21. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From study start to end of Primary Phase (Study Day 245)
Population: The analysis was based on the ITT population, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 34 | 17 | 12
Participants | 1 | 0 | 0

22. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 21
Time Frame: During the entire study period (Up to Day 105 of Booster Phase)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
Number analyzed (Participants) | 34 | 17 | 12
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: within 7 days (Days 0-6) post-orimary vaccination. Unsolicited adverse events (AEs): within 30 days (Days 0-29) post-primary vaccination and post-CHMI. Serious adverse events (SAEs): during the entire study period (up to Day 105 of Booster Phase).
Description: Solicited and Unsolicited results were not reported for the Infectivity Control Group, since subjects from this group did not receive any immunization.
Arm/Group | GSK257049-0,1,7M Group | GSK257049-0,1,2M Group | Infectivity Control Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/17 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/17 | 0/12
Other Adverse Events (participants affected / at risk) | 34/34 | 17/17 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK257049-0,1,7M Group (N=34) | GSK257049-0,1,2M Group (N=17) | Infectivity Control Group (N=12)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK257049-0,1,7M Group (N=34) | GSK257049-0,1,2M Group (N=17) | Infectivity Control Group (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0
Arthropod bite (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0
Chills (General disorders) | 4 (5) | 4 (5) | 0
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0
Erythema (Skin and subcutaneous tissue disorders) | 27 (50) | 13 (23) | 0
Fatigue (General disorders) | 20 (39) | 10 (19) | 0
Feeling hot (General disorders) | 3 (3) | 2 (2) | 0
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 8 (15) | 8 (12) | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0
Headache (Nervous system disorders) | 21 (44) | 12 (30) | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 4 (6) | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0
Pain (General disorders) | 32 (88) | 16 (43) | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0
Pyrexia (General disorders) | 8 (9) | 4 (4) | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0
Swelling (General disorders) | 23 (39) | 6 (8) | 0
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 7 (7) | 0
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.